CLINICAL TRIAL: NCT07307326
Title: An Examination of the Feasibility of a Brief Personalized Alcohol Biomarker Feedback Intervention for High-risk College Students
Brief Title: Biomarker Feedback Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kimberly Mallett, Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00027939
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: High Risk Drinking; College Student Drinking
Keywords: college student drinking
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: The first group receives the e-CTG + TAC feedback and the second group receives the e-CTG-only.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCHECKUP TO GO (eCTG) (Experimental): A brief, web-based program designed by San Diego State University to reduce high-risk drinking by providing personalized normative feedback regarding alcohol use, risk factors, and risks associated with drinking and accurate information about alcohol
  Interventions: Behavioral: eCHECKUP TO GO (eCTG)
- eCHECKUPTOGO + brief personalized biomarker feedback intervention (eCTG + TAC) (Experimental): Participants will receive the eCHECKUPTOGO in addition to the transdermal alcohol concentration (TAC) personalized feedback. The TAC is a brief individually delivered intervention based on the principles of Motivational Interviewing and focuses on increasing students' motivation to reduce harmful drinking by drinking in a safer, less risky manner. Participants will receive information on their drinking (both from the TAC sensor and daily diary data). Participants will be asked about drinking events during the past 2 weeks (how reflective they were of typical patterns and if a night stood out as particularly negative). Students will receive information and visual representations about TAC rise rates and peaks, and then be shown how their drinking during the past 2 weeks maps onto those visuals.
  Interventions: Behavioral: eCHECKUPTOGO + brief personalized alcohol biomarker feedback intervention (eCTG + TAC)

INTERVENTIONS:
Behavioral: eCHECKUP TO GO (eCTG) — A brief, web-based program designed by San Diego State University to reduce high-risk drinking by providing personalized normative feedback regarding alcohol use, risk factors, and risks associated with drinking and accurate information about alcohol
  Arms: eCHECKUP TO GO (eCTG)
Behavioral: eCHECKUPTOGO + brief personalized alcohol biomarker feedback intervention (eCTG + TAC) — Participants will receive the eCHECKUPTOGO in addition to the transdermal alcohol concentration (TAC) personalized feedback. The TAC is a brief individually delivered intervention based on the principles of Motivational Interviewing and focuses on increasing students' motivation to reduce harmful drinking by drinking in a safer, less risky manner. Participants will receive information on their drinking (both from the TAC sensor and daily diary data). Participants will be asked about drinking events during the past 2 weeks (how reflective they were of typical patterns and if a night stood out as particularly negative). Students will receive information and visual representations about TAC rise rates and peaks, and then be shown how their drinking during the past 2 weeks maps onto those visuals.
  Arms: eCHECKUPTOGO + brief personalized biomarker feedback intervention (eCTG + TAC)

SUMMARY:
The goal of the study is to examine alcohol use behaviors of young adults through the use of testing the feasibility of adding an innovative brief personalized alcohol biomarker feedback component (TAC feedback) to an existing efficacious personalized feedback intervention, eCHECKUP TO GO (eCTG), and how (if at all) the intervention impacts drinking behaviors in high-risk college students. The study will conduct a feasibility assessment of the TAC feedback component, and will also assess the effects of the eCTG + TAC at 6-months post-baseline relative to an eCTG only group.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-23 at enrollment
* Endorse drinking 4+/5+ (women/men) on a typical Friday or Saturday in the past 3-months
* Report at least 1 alcohol-induced blackout in the past 3-months
* Willing to wear a TAC sensor for 14 days at Waves 1 and 2

Exclusion Criteria:

* Younger than 18 at baseline
* Not fluent in English
* No Internet access

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Examine changes in Transdermal Alcohol Concentration (TAC) rise rate | Baseline, 6 months
  TAC rise rate will be collected via the BACtrack Skyn wrist sensor, which measures transdermal alcohol concentration (TAC) in micrograms of ethanol per liter of air every 20 seconds to obtain biomarkers - rise rate is a TAC increase.
Examine changes in Transdermal Alcohol Concentration (TAC) peak intoxication level | Baseline, 6 months
  TAC peak will be collected via the BACtrack Skyn wrist sensor, which measures transdermal alcohol concentration (TAC) in micrograms of ethanol per liter of air every 20 seconds to obtain biomarkers - peak is the maximum TAC recorded per day.
Examine high risk drinking days | Baseline, 6 months
  Heavy episodic drinking (HED) days are recorded when women indicate drinking 4+ drinks in 2 hour window/men indicate drinking 5+ drinks in 2 hour window. High-intensity drinking (HID) days are recorded when women indicate drinking 8+ drinks in 2 hour window/men indicate drinking 10+ drinks in 2 hour window.

SECONDARY OUTCOMES:
Examine negative consequences of alcohol use | Baseline, 6 months
  Alcohol related consequences (e.g., said or done embarrassing things) from the past 3 months will be measured using the established Brief Young Adult Alcohol Consequences Questionnaire. Response options will be on a 5-point scale ranging from (0) No or not in the past 3 months to (4) 4 or more times. Consequences will also be measures during the daily surveys on a Yes/No response scale.
Examine Alcohol Use Disorder (AUD) symptoms | Baseline, 6 months
  Alcohol use disorder symptoms will be measured using the Alcohol Use Disorder Module of the SCID-5 and will be via in-person interview at baseline (past 12-months) and 6-month (past 6-months).

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Mallett, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of funding requirements, data collected will be submitted to the NIAAA Data Archive.
Access Criteria: Individuals will request access to the data via a data access request through the data archive.